CLINICAL TRIAL: NCT06182033
Title: Penetrating the Classroom Social Network for Children With Language Impairment Via Peer Mediated Intervention
Acronym: PEERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R21DC018395 (NIH)
Record Dates: First submitted 2023-12-04; First posted 2023-12-26 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Peer Influence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-mediated pivotal response intervention (Experimental): Facilitators hold four 15-minute training sessions with the peer group to engage the target child. The facilitator explicitly identifies the "buddy" and asks the children to use four strategies to play with the child during center time: (a) offer your buddy some play options; (b) show and talk about how to play with your buddy; (c) compliment your buddy; and (d) show your buddy how to take turns. At each training session the facilitator will describe one strategy, provide examples, and practice the strategy through role play. After trainings, the facilitator provides ongoing support during center time to implement the strategies over 12 weeks during months 3-6 of the 9 months of study participation.
  Interventions: Behavioral: Peer-mediated pivotal response training
- Control (No Intervention): Business as usual

INTERVENTIONS:
Behavioral: Peer-mediated pivotal response training — Teachers support children in the implementation of three strategies directed toward a target child identified as having language impairment and as isolated from the classroom social network.
  Arms: Peer-mediated pivotal response intervention

SUMMARY:
This exploratory experiment is designed to determine the extent to which the socialization experiences and social, behavioral, and linguistic skills of preschoolers with language impairment (LI) can be improved. The investigators implement a peer-mediated intervention in inclusive preschool classrooms, randomly assigned to treatment (n=12) or control (n=13) conditions. A focal child is identified in each classroom, representing a child with LI (3 to 5 years of age) who exhibits the poorest pragmatic-language skills and highest level of social exclusion in the classroom. Over a 12-week period, the focal children will receive peer-mediated intervention from identified peers, who use strategies to engage the focal child socially during center time, as supported by a classroom facilitator (teacher, aide). Outcomes of interest include the overarching classroom social network and its embedded socialization processes (e.g., frequency of child-to-child interaction), the focal child's interactions with peers and exposure to peer talk, and the focal child's social, behavioral, and linguistic skills. The study employs state-of-the-art social network analyses to represent the classroom network at the child, dyad, and network level and is dynamically modeled over the academic year using advanced location-tracking technologies and voice-activated recorders to capture incoming and outgoing peer talk for the focal child. The investigators anticipate the results of this study to yield significant theoretical and scientific impact. Theoretically, the investigators propose that improved socialization experiences in the preschool classroom can disrupt the social exclusion and peer maltreatment experienced by children with LI, leading to accelerated growth in linguistic, social, and behavioral outcomes for children with LI.

DETAILED DESCRIPTION:
This study involves 25 inclusive preschool classrooms. The study uses an randomized controlled trial to estimate treatment impacts of a peer-mediated intervention, with 12 classrooms assigned to the treatment condition and 13 to the control condition. Within each classroom, the focal participants are children isolated from their classroom social network with low pragmatic language skills. One target child is selected per classroom using a priori exclusionary and inclusionary criteria. In the fall of each year, simple random assignment is used to allocate classrooms to the treatment group and to the control group. First, investigators identify all children's positions within the classroom social network using a teacher matrix conducted in fall of the academic year; from this network a child-level social network index is calculated (i.e., individual degree centrality; lower scores are characteristic of social exclusion). Second, teachers simultaneously complete the Developmental Pragmatic Profile (DPP) for each child in the classroom. Finally, among the participating focal children, investigators select the target child based on the lowest centrality scored weighted by DPP score, so that focal children represent the most socially isolated children with the poorest social-pragmatic communication skills. Children and teachers participate for a 9-month period, and the primary approach to treatment for focal children is described here. Specifically, focal children in classrooms randomized to the treatment condition receive peer-mediated pivotal response training (PRT) per procedures detailed by Brock et al.. PRT procedures are facilitated by a classroom facilitator-a classroom teacher or teaching assistant-who receives ongoing training and support from research staff.

First, investigators provide a one-on-one 1-h training session for each facilitator that focuses on how to identify, initially train, and then support peers on a day-to-day basis during center time. Second, investigators partner with the facilitator to identify two peers who (a) demonstrate good social skills; (b) respond well to adult directions; (c) have consistent attendance; and (d) do not have a history of negative interactions with the target student. The facilitator explicitly identifies the focal child ("buddy") and asks the children to use three strategies to play with the buddy during center time: (a) offer buddy some play options; (b) show and talk about how to play with buddy; (c) compliment buddy. At each training session the facilitator describes one strategy, provides examples, and has peers practice the strategy through role play. During the role play the facilitator encourages and coaches peers to use the strategy as intended. The facilitator then provides ongoing support to peers during center time to implement the strategies by helping peers to set goals immediately before center time for use of the strategies, regularly encouraging peers and supporting peers to use the strategies, praising peers for use of the strategies, and reviewing peers' goals and interactions with the focal child at the end of center time. Facilitators provide this support during center time at least three times weekly for a 12-week period. The investigators propose that improved socialization experiences in the preschool classroom for focal children can disrupt the social exclusion, leading to accelerated growth in linguistic, social, and behavioral outcomes.

ELIGIBILITY:
General Inclusion Criteria

* teacher informed consent
* caregiver informed consent
* 36 months of age or older.

Exclusion Criteria:

* no caregiver informed consent
* younger than 36 months of age

Ages: 36 Months to 66 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Justice, PhD, Principal Investigator — Ohio State University
Locations (1):
- Crane Center for Early Childhood Research and Policy, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foster TJ, Xiao N, Pelfrey GL, Villasanti HG, Brock M, Justice L. Peer-Mediated Intervention for Socially Isolated Preschoolers: An Early-Stage Feasibility Study. Lang Speech Hear Serv Sch. 2024 Jan 11;55(1):166-180. doi: 10.1044/2023_LSHSS-23-00090. Epub 2023 Dec 4. PMID 38048318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Classrooms were randomly assigned to condition. One target child was selected within each classroom prior to random assignment. As such, the number of classrooms in the study and the number of target children analyzed and reported are equivalent. Target children in classrooms assigned to the treatment condition experienced peer-mediated pivotal response training. Target children in control classrooms experiences business as usual.
Units Other Than Participants: classrooms
Period: Overall Study
Arm/Group | Peer-mediated Pivotal Response Intervention | Control
Started | 15; 15 classrooms | 15; 15 classrooms
Baseline Assessments | 14; 14 classrooms | 14; 14 classrooms
Timepoint 2 Assessment | 12; 12 classrooms | 13; 13 classrooms
Completed | 12; 12 classrooms | 13; 13 classrooms
Not Completed | 3; 3 classrooms | 2; 2 classrooms
Not completed — No baseline survey provided. Needed for target child selection. | 1 | 1
Not completed — Target child relocation | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: This excludes children who attrited from the project as summarized in the participant flow section of this report.
Groups:
- Peer Mediated Pivotal Response Intervention: Facilitators hold four 15-minute training sessions with the peer group to engage the target child. The facilitator explicitly identifies the "buddy" and asks the children to use four strategies to play with the child during center time: (a) offer your buddy some play options; (b) show and talk about how to play with your buddy; (c) compliment your buddy; and (d) show your buddy how to take turns. At each training session the facilitator will describe one strategy, provide examples, and practice the strategy through role play. After trainings, the facilitator provides ongoing support during center time to implement the strategies over 12 weeks during months 3-6 of the 9 months of study participation.
  Peer-mediated pivotal response training: Teachers support children in the implementation of three strategies directed toward a target child identified as having language impairment and as isolated from the classroom social network
- Total: Total of all reporting groups
Arm/Group | Peer Mediated Pivotal Response Intervention | Control | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: months] | 50.42 (8.37) | 51.77 (11.04) | 51.12 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 8 | 10 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity: Black non-hispanic | 1 | 2 | 3
  Race and Ethnicity: White non-Hispanic | 6 | 10 | 16
  Race and Ethnicity: Hispanic | 2 | 0 | 2
  Race and Ethnicity: Multiracial-non-Hispanic | 0 | 1 | 1
  Race and Ethnicity: Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 13 | 25
Preschool Language Screener 5 GROWTH SCALE VALUE [Mean (Standard Deviation); unit: Score on a scale] — The PLS-5 is used to assess expressive language skills. Specific skills assessed include naming, expressing quantity, describing, using specific prepositions, grammatical markers, sentence structures, and emergent literacy skills. An assessor indicates whether a child passes (1) or does not pass (0) each item. Growth Scale Value: Range: Minimum = 100/Max = 900. Higher scores indicate better expressive language skills. Assessed at baseline, 3 months, and 9 months. Baseline reported.
  Score on a scale | 437.09 (38.55) | 455.38 (53.40) | 447 (47.12)

OUTCOME MEASURES:

1. Primary Outcome: Preschool Language Screener 5 (PLS-5) - Growth Scale Value
Description: The PLS-5 is used to assess expressive language skills. Specific skills assessed include naming, expressing quantity, describing, using specific prepositions, grammatical markers, sentence structures, and emergent literacy skills. An assessor indicates whether a child passes (1) or does not pass (0) each item. Growth Scale Value: Range: Minimum = 100/Max = 900. Higher scores indicate better expressive language skills. Assessed at baseline, 3 months, and 9 months. Baseline reported.
Time Frame: at baseline, 3 months, and 9 months
Population: At baseline and 3 months, 11 participants were assessed with the PLS-5 in the peer-mediated pivotal response intervention group instead of the total number in the sample (n = 12) because one participant was consistently absent from school during the assessment window. At 9 months, 12 participants were assessed with the PLS-5 in the control group instead of the total number in the sample (n = 13) because one participant was consistently absent from school during the assessment window.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer-mediated Pivotal Response Intervention | Control
Number analyzed (Participants) | 12 | 13
score on a scale
  Baseline: number analyzed (Participants) | 11 | 13
  Baseline | 437.09 (38.55) | 455.38 (53.40)
  3 months: number analyzed (Participants) | 11 | 13
  3 months | 459.09 (40.59) | 464.77 (52.32)
  9 months: number analyzed (Participants) | 12 | 12
  9 months | 459.08 (36.59) | 478.58 (42.37)
Statistical Analysis 1: Comparison: Peer-mediated Pivotal Response Intervention vs Control; We conducted a linear regression. We accounted for baseline, which allowed us to examine residualized gains. We controlled for age; Test type: Other; p = .84, Regression, Linear; Kenward Rogers and Restricted Maximum Likelihood adjustment made to reduce error likelihood

2. Secondary Outcome: Developmental Pragmatic Profile (DPP)
Description: A 26-item psychometrically sound checklist assessing children's pragmatic skills (e.g., conversational abilities, giving information), and DPP scores have strong classification accuracy in differentiating children with LI from non-affected classmates. This profile identifies non-verbal and verbal pragmatic deficits that may negatively influence social and academic communication in context. The questionnaire uses a 1 (never) to 4 (always) rating scale to assess the child's ability to appropriately communicate in social situations (i.e., "communicates [verbally and nonverbally] when playing with other children" or "introduces new conversation topics"). There is also a Not Appropriate option which indicates that the items is "Not appropriate for the child (culturally or other reason)." Raw Score Range: Minimum = 26/Max = 104. Higher scores on the DPP indicate greater language skills. Raw score is calculated by summing scores across the 26 items comprising the DPP.
Time Frame: at baseline and 9 months, month 9 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer-mediated Pivotal Response Intervention | Control
Number analyzed (Participants) | 12 | 13
score on a scale | 68.75 (18.54) | 77.42 (12.46)
Statistical Analysis 1: Comparison: Peer-mediated Pivotal Response Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = .727, Regression, Linear; Kenward Rogers and Restricted Maximum Likelihood adjustment made to reduce error likelihood

3. Secondary Outcome: Teacher-Child Rating Scale (TCRS)
Description: The Teacher-Child Rating Scale is a 32-item teacher-report instrument that measures children's social competence. Teachers respond to statements on a 5-point scale (1 = strongly disagree, 5 = strongly agree). To calculate each subscale score, one must sum positive items; sum negative items; subtract the sum of negative times from the number 24; sum this value with the sum of the positive items.
  Assertiveness Subscale: Range: (Min: 8/Max: 40 ) Behavior Control Subscale: (Min: 8/Max: 40) Peer Social Skills Subscale: (Min: 8/Max: 40) Talk Orientation Subscale: (Min: 8/Max: 40)
  Higher scores indicate higher skills as measured by each subscale.
Time Frame: at baseline, and 9 months, month 9 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer-mediated Pivotal Response Intervention | Control
Number analyzed (Participants) | 12 | 13
score on a scale
  Assertiveness | 25.50 (5.89) | 28.42 (7.04)
  Behavior Control | 25.42 (7.85) | 26.67 (7.45)
  Peer Social Skills | 26 (10.22) | 27.25 (7.84)
  Task Orientation | 25 (6.09) | 26.5 (9.15)
Statistical Analysis 1: Comparison: Peer-mediated Pivotal Response Intervention vs Control; These analyses use the assertiveness subscale as the outcome variable. We conducted a linear regression for each of the measure's subscales. We accounted for baseline, which allowed us to examine residualized gains. We controlled for age; Test type: Other; p = .205, Regression, Linear; Kenward Rogers and Restricted Maximum Likelihood adjustment made to reduce error likelihood
Statistical Analysis 2: Comparison: Peer-mediated Pivotal Response Intervention vs Control; This analysis focused specifically on the behavior control subscale. We conducted a linear regression for each of the measure's subscales. We accounted for baseline, which allowed us to examine residualized gains. We controlled for age; Test type: Other; p = .034, Regression, Linear; Kenward Rogers and Restricted Maximum Likelihood adjustment made to reduce error likelihood
Statistical Analysis 3: Comparison: Peer-mediated Pivotal Response Intervention vs Control; These analyses use the Task Orientation subscale as the outcome variable. We conducted a linear regression for each of the measure's subscales. We accounted for baseline, which allowed us to examine residualized gains. We controlled for age; Test type: Other; p = .099, Regression, Linear; Kenward Rogers and Restricted Maximum Likelihood adjustment made to reduce error likelihood
Statistical Analysis 4: Comparison: Peer-mediated Pivotal Response Intervention vs Control; This analysis used peer social skills subscale as the outcome in the model. We conducted a linear regression for each of the measure's subscales. We accounted for baseline, which allowed us to examine residualized gains. We controlled for age; Test type: Other; p = .209, Regression, Linear

4. Secondary Outcome: Peer Incoming Talk
Description: Researchers record the amount of incoming talk focal children experience using a hands-free voice-activated recorder worn by the child, with audio capture transcending the entire classroom day. Investigators process these recordings to capture incoming talk with proximate peers using the following process: (i) augment the voice-recorder ability/voice detection/processing algorithms from the Matlab Audio Systems Toolbox to determine if people are speaking; and (i) use 2D-proximity data from continuous location tracking to parse the audio into the cases where there is simultaneous peer proximity and recorded voice. Incoming peer talk will be used to calculated in-degree centrality for each child on each of 8 randomly selected recording days to examine change in in-degree centrality over the course of an academic year. Talk is operationalized as utterances per minute. An utterance is a continuous piece of speech by an individual before or after which there is silence.
Time Frame: through study completion, an average of 9 months, month 9 reported
Measure: Mean (Standard Deviation); unit: utterances per minute--final observation
Arm/Group | Peer-mediated Pivotal Response Intervention | Control
Number analyzed (Participants) | 12 | 13
utterances per minute--final observation | 5.86 (5.41) | 6.35 (4.35)
Statistical Analysis 1: Comparison: Peer-mediated Pivotal Response Intervention vs Control; We examined the trajectory across timepoints using a multilevel model that controlled for age. The p value is in reference to the difference between the treatment and control children at the final observation; Test type: Other; p = .82, Multilevel Model; Kenward Rogers and Restricted Maximum Likelihood adjustment made to reduce error likelihood

5. Secondary Outcome: Peer Outgoing Talk
Description: Researchers record the amount of outgoing talk vocalized by focal children using a hands-free voice-activated recorder worn by the child, with audio capture transcending the entire classroom day. Investigators process these recordings to capture incoming talk with proximate peers using the following process: (i) augment the voice-recorder ability/voice detection/processing algorithms from the Matlab Audio Systems Toolbox to determine if people are speaking; and (i) use 2D-proximity data from continuous location tracking to parse the audio into the cases where there is simultaneous peer proximity and recorded voice. Incoming peer talk will be used to calculated out-degree centrality for each child on each of 8 randomly selected recording days to examine change in out-degree centrality over the course of an academic year. Talk is operationalized as utterances per minute. An utterance is a continuous piece of speech by an individual before or after which there is silence.
Time Frame: through study completion, an average of 9 months, month 9 reported
Measure: Mean (Standard Deviation); unit: outgoing utterances per minute-final obs
Arm/Group | Peer-mediated Pivotal Response Intervention | Control
Number analyzed (Participants) | 12 | 13
outgoing utterances per minute-final obs | 4.68 (11.34) | 5.22 (3.73)
Statistical Analysis 1: Comparison: Peer-mediated Pivotal Response Intervention vs Control; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = .67, Multilevel Model; Kenward-Rogers and Restricted Maximum Likelihood adjustments in light of small sample size to reduce error likelihood

6. Secondary Outcome: Peer Interactions
Description: Peer interactions of focal children were observed 4 times over the academic year using Brock's established protocol. Researchers observe the focal child for 30 minutes during center time and apply a partial interval recording system involving 15 s of observation and 45 s of documentation. For peer interactions, each interval is coded for whether the target child is interacting with peers. These observation data will be used to calculate frequency of peer interactions experienced by target children during the 30-minute observation. Reliability will be assessed for 20% of observations via double-coding with observers blind to classroom and child condition.
Time Frame: through study completion, an average of 9 months, final observation (up to 9 months) reported
Measure: Mean (Standard Deviation); unit: percentage of intervals
Arm/Group | Peer-mediated Pivotal Response Intervention | Control
Number analyzed (Participants) | 12 | 13
percentage of intervals
  Incoming Peer Interactions | 43 (15.9) | 21.7 (19.6)
  Outgoing Peer Interactions | 42.3 (18.4) | 22 (17.4)
Statistical Analysis 1: Comparison: Peer-mediated Pivotal Response Intervention vs Control; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = .024, Regression, Linear; Kenward-Rogers and Restricted Maximum Likelihood to account for the small sample size

7. Secondary Outcome: Play Interactions
Description: Play interactions of focal children will be observed 4 times over the academic year using Brock's established protocol. Observers will observe the focal child for 30 minutes during center time and apply a partial interval recording system involving 15 s of observation and 45 s of documentation. For play interactions, each interval is coded for whether the target child is engaged in play with peers. These observation data will be used to calculate frequency of play interactions experienced by target children during the 30-minute observation. Reliability will be assessed for 20% of observations via double-coding with observers blind to classroom and child condition.
Time Frame: through study completion, an average of 9 months; final observation (up to 9 months) reported
Measure: Mean (Standard Deviation); unit: percentage of intervals
Arm/Group | Peer-mediated Pivotal Response Intervention | Control
Number analyzed (Participants) | 12 | 13
percentage of intervals | 43 (25.9) | 24.7 (23.1)
Statistical Analysis 1: Comparison: Peer-mediated Pivotal Response Intervention vs Control; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = .013, Regression, Linear; Kenward Rogers and Restricted Maximum Likelihood adjustment made to reduce error likelihood

ADVERSE EVENTS:
Time Frame: No formal monitoring occurred. Researchers interacted with participants over the 9-month period of their study involvement.
Description: All cause mortality and serious adverse events were not formally monitored. No drugs or medical procedures were administered to subjects as part of this study. The research activities reported herein were deemed as minimal risk by the Institutional Review Board responsible for the oversight of this study. No adverse events occurred throughout the duration of the project. Study activities were monitored by checking in with research partners when visiting schools for data collection.
Groups:
- Peer-mediated Pivotal Response Training: Facilitators hold four 15-minute training sessions with the peer group to engage the target child. The facilitator explicitly identifies the "buddy" and asks the children to use four strategies to play with the child during center time: (a) offer your buddy some play options; (b) show and talk about how to play with your buddy; (c) compliment your buddy; and (d) show your buddy how to take turns. At each training session the facilitator will describe one strategy, provide examples, and practice the strategy through role play. After trainings, the facilitator provides ongoing support during center time to implement the strategies over 12 weeks during months 3-6 of the 9 months of study participation.
Arm/Group | Peer-mediated Pivotal Response Training | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13

LIMITATIONS AND CAVEATS:
The study protocol initially included the use of a waitlist control design. Given the study pause due to the impacts of the global pandemic and the landscape of early childhood education centers in the subsequent years during which study activities were implemented, our team instead opted to randomly assign participating classrooms to a study condition in lieu of the waitlist control design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT06182033/Prot_SAP_000.pdf